CLINICAL TRIAL: NCT01832480
Title: Trichomonas Vaginalis Repeat Infections Among HIV Negative Women
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tulane University Health Sciences Center (Other)
Responsible Party: Principal Investigator, Patricia Kissinger, Professor, Tulane University Health Sciences Center
Organization: Tulane University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4042013
Record Dates: First submitted 2013-04-04; First posted 2013-04-16 (Estimated); Results first posted 2019-02-12 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2019-01

CONDITIONS: Vaginitis Trichomonal or Due to Trichomonas
Keywords: Trichomonas vaginalis; metronidazole
MeSH Terms: conditions — Trichomonas Vaginitis

STUDY DESIGN:
Masking Description: This was an open label study
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MTZ 2 g (Active Comparator): Single dose MTZ
  Interventions: Drug: MTZ 2 g
- MTZ 500 mg twice daily x 7 days (Experimental): Multi dose MTZ
  Interventions: Drug: MTZ 500 mg twice daily x 7 days

INTERVENTIONS:
Drug: MTZ 500 mg twice daily x 7 days — MTZ 500 mg twice daily x 7 days
  Other Names: Multi-dose MTZ
  Arms: MTZ 500 mg twice daily x 7 days
Drug: MTZ 2 g — MTZ 2 g
  Other Names: Single dose MTZ
  Arms: MTZ 2 g

SUMMARY:
The overall goal of this project is to determine the influence of patient treatment and host factors on repeat Trichomonas vaginalis (TV) infections among HIV-negative women

DETAILED DESCRIPTION:
This study is a phase III randomized clinical trial. HIV-negative women who test positive for TV at their routine gynecological exam at participating clinics will be referred to the nurse/study coordinator to screen for eligibility, provide a description of the study, and obtain written, informed consent (N=700). Subjects will undergo an audio computer assisted self- interview (ACASI), and will self-collect vaginal swabs for Trichomonas testing by InPouch and Nucleic Acid Amplification Test (NAAT), Gram stain testing, and a future microbiome specimen. They will be randomized into one of two arms; metronidazole (MTZ) 2 g single dose (CDC recommended treatment regimen) or MTZ 500 mg twice daily x 7-day dose (CDC alternative treatment regimen). All enrolled women will be scheduled for a follow-up visit at four weeks post treatment completion (window 3-13 weeks).

ELIGIBILITY:
Inclusion Criteria:

* female
* English speaking
* >= 18 years old

Exclusion Criteria:

* HIV-infected
* unable to provide informed consent
* pregnant
* breast feeding
* treated by their provider for Bacterial vaginosis (BV) at visit

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 623 (Actual)
Dates: Start 2014-10-06 (Actual); Primary Completion 2017-06-05 (Actual); Study Completion 2017-06-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Kissinger, MD, Principal Investigator — Tulane Univeristy
Locations (3):
- United States (3):
  - Jefferson County Dept of Health/STD Specialty Clinic, Birmingham, Alabama
  - CrescentCare Health and Wellness Center, New Orleans, Louisiana
  - Crossroads Clinic, Jackson, Mississippi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kissinger P, Amedee A, Clark RA, Dumestre J, Theall KP, Myers L, Hagensee ME, Farley TA, Martin DH. Trichomonas vaginalis treatment reduces vaginal HIV-1 shedding. Sex Transm Dis. 2009 Jan;36(1):11-6. doi: 10.1097/OLQ.0b013e318186decf. PMID 19008776
- [Background] Kissinger P, Secor WE, Leichliter JS, Clark RA, Schmidt N, Curtin E, Martin DH. Early repeated infections with Trichomonas vaginalis among HIV-positive and HIV-negative women. Clin Infect Dis. 2008 Apr 1;46(7):994-9. doi: 10.1086/529149. PMID 18444815
- [Background] Kissinger P, Schmidt N, Mohammed H, Leichliter JS, Gift TL, Meadors B, Sanders C, Farley TA. Patient-delivered partner treatment for Trichomonas vaginalis infection: a randomized controlled trial. Sex Transm Dis. 2006 Jul;33(7):445-50. doi: 10.1097/01.olq.0000204511.84485.4c. PMID 16531939
- [Background] Kissinger P, Mena L, Levison J, Clark RA, Gatski M, Henderson H, Schmidt N, Rosenthal SL, Myers L, Martin DH. A randomized treatment trial: single versus 7-day dose of metronidazole for the treatment of Trichomonas vaginalis among HIV-infected women. J Acquir Immune Defic Syndr. 2010 Dec 15;55(5):565-71. doi: 10.1097/QAI.0b013e3181eda955. PMID 21423852
- [Background] Howe K, Kissinger PJ. Single-Dose Compared With Multidose Metronidazole for the Treatment of Trichomoniasis in Women: A Meta-Analysis. Sex Transm Dis. 2017 Jan;44(1):29-34. doi: 10.1097/OLQ.0000000000000537. PMID 27898571
- [Background] Meites E, Gaydos CA, Hobbs MM, Kissinger P, Nyirjesy P, Schwebke JR, Secor WE, Sobel JD, Workowski KA. A Review of Evidence-Based Care of Symptomatic Trichomoniasis and Asymptomatic Trichomonas vaginalis Infections. Clin Infect Dis. 2015 Dec 15;61 Suppl 8(Suppl 8):S837-48. doi: 10.1093/cid/civ738. PMID 26602621
- [Background] Kissinger P. Trichomonas vaginalis: a review of epidemiologic, clinical and treatment issues. BMC Infect Dis. 2015 Aug 5;15:307. doi: 10.1186/s12879-015-1055-0. PMID 26242185

RESULTS

PARTICIPANT FLOW:
Groups:
- Metronidazole (MTZ) 2 g: Single dose MTZ
  MTZ 2 g: MTZ 2 g
- Metronidazole (MTZ) 500 mg Twice Daily x 7 Days: Multi dose MTZ
  MTZ 500 mg twice daily x 7 days
Period: Overall Study
Arm/Group | Metronidazole (MTZ) 2 g | Metronidazole (MTZ) 500 mg Twice Daily x 7 Days
Started | 311 | 312
Completed | 270 | 270
Not Completed | 41 | 42
Not completed — Lost to Follow-up | 33 | 30
Not completed — Withdrawal by Subject | 0 | 2
Not completed — post randomization ineligible | 8 | 10

BASELINE CHARACTERISTICS:
Groups:
- Metronidazole (MTZ) 500 mg BID x 7 Days: Multi dose MTZ
  MTZ 500 mg BID x 7 days: MTZ 500 mg BID x 7days
- Total: Total of all reporting groups
Arm/Group | Metronidazole (MTZ) 2 g | Metronidazole (MTZ) 500 mg BID x 7 Days | Total
Number analyzed (Participants) | 311 | 312 | 623
Age, Customized [Count of Participants; unit: Participants] — Population: there were 3 subjects with missing age.
  Participants
    >=30 years: number analyzed (Participants) | 309 | 310 | 619
    >=30 years | 132 | 116 | 248
    <30 years | 178 | 193 | 371
    missing | 2 | 1 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 311 | 312 | 623
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 293 | 298 | 591
  White | 12 | 8 | 20
  More than one race | 4 | 4 | 8
  Unknown or Not Reported | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 311 | 312 | 623

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects That Were Trichomonas Vaginalis (TV) Positive After Treatment With Metronidazole (MTZ)
Description: Presence of TV is assessed by nucleic acid amplification test (NAAT) of vaginal swab collected 4 weeks post treatment completion.
Time Frame: 4 weeks post treatment completion
Population: 570 cases available. Multiple imputation performed for those with missing Test of Cure (TOC) data.
Measure: Count of Participants; unit: Participants
Groups:
- Trichomonas (TV) Positive After 2 g Dose: Subjects who were randomized to MTZ singe dose (2g) and tested TV positive at test of cure
- Trichomonas (TV) Positive After Metronidazole (MTZ) Multi Dose: Subjects who were randomized to MTZ multi dose (500mg twice daily x 7 days) and tested TV positive at test of cure
Arm/Group | Trichomonas (TV) Positive After 2 g Dose | Trichomonas (TV) Positive After Metronidazole (MTZ) Multi Dose
Number analyzed (Participants) | 311 | 312
Participants | 58 | 34

ADVERSE EVENTS:
Time Frame: 4 weeks post completion of treatment
Description: A standard event reporting form will be used by all sites. In the event of an adverse event, the form was filled out by study personnel within 24 hours of the reporting of the event and sent to the investigators for review.
Groups:
- Metronidazole (MTZ) 2 g: This is the control dose arm.
- Metronidazole (MTZ) 500 mg Twice Daily x 7 Days Dose: This is the experimental dose arm.
Arm/Group | Metronidazole (MTZ) 2 g | Metronidazole (MTZ) 500 mg Twice Daily x 7 Days Dose
All-Cause Mortality (participants affected / at risk) | 0/311 | 0/312
Serious Adverse Events (participants affected / at risk) | 0/311 | 2/312
Other Adverse Events (participants affected / at risk) | 90/311 | 89/312
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metronidazole (MTZ) 2 g (N=311) | Metronidazole (MTZ) 500 mg Twice Daily x 7 Days Dose (N=312)
spontaneous abortion (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 2 (2) — women tested negative for pregnancy at baseline but were found to be pregnant at follow-up and had a spontaneous abortion that may or may not have been a results of the medication
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metronidazole (MTZ) 2 g (N=311) | Metronidazole (MTZ) 500 mg Twice Daily x 7 Days Dose (N=312)
nausea (Gastrointestinal disorders) | 61 (61) | 63 (63)
headache (Nervous system disorders) | 15 (15) | 24 (24)
Vomiting (Gastrointestinal disorders) | 7 (7) | 13 (13)
Dizziness (Nervous system disorders) | 18 (18) | 16 (16)
Bad taste in mouth (General disorders) | 6 (6) | 4 (4)
Vaginal itching (Reproductive system and breast disorders) | 1 (1) | 3 (3)
Fatigue (General disorders) | 3 (3) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Yeast infections (Reproductive system and breast disorders) | 1 (1) | 2 (2)
Stomach Pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Verbal intimidation by partner (General disorders) | 1 (1) | 1 (1)
Vision change (Eye disorders) | 1 (1) | 0 (0)
Persistent nausea/vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) — This was recorded as a single adverse event
Increased bowel movements (Gastrointestinal disorders) | 0 (0) | 1 (1)
Numbness (Nervous system disorders) | 1 (1) | 1 (1)
Restlessness (General disorders) | 0 (0) | 1 (1)
Vaginal bleeding (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Loss of appetite (General disorders) | 1 (1) | 0 (0)
Depression (General disorders) | 1 (1) | 1 (1) — Not clinically assessed, described as feeling low
Gas (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hot flashes (General disorders) | 1 (1) | 0 (0)
General feeling sick (General disorders) | 0 (0) | 1 (1)
Dry mouth (General disorders) | 0 (0) | 1 (1)
Dark urine (Renal and urinary disorders) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Peeling skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Myalagia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Altered mental state (General disorders) | 1 (1) | 0 (0)
Stiff neck (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-02): https://cdn.clinicaltrials.gov/large-docs/80/NCT01832480/Prot_SAP_000.pdf